CLINICAL TRIAL: NCT02325245
Title: Randomized-Controlled Trial of Metformin to Prevent Frailty in Pre-frail Elderly
Brief Title: Effects of Metformin in Pre-frail Elderly
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Purwita Wijaya Laksmi, Purwita Wijaya Laksmi, MD, SpPD-KGer, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FRAIL-01
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Pre-frail Elderly
Keywords: Frailty; Pre-frailty; Metformin; Elderly; Quality of life; Handgrip; Gait speed; Myostatin
MeSH Terms: conditions — Frailty | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): Metformin tablet 500 mg three times a day for 16 weeks.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo tablet three times a day for 16 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin tablet 500 mg three times a day for 16 weeks. If there is no significant outcome obtained between two arms in 16 weeks, metformin will continue until 24 weeks.
  Other Names: CAS Number: 657-24-9; ATC Code: A10BA02
  Arms: Metformin
Drug: Placebo — Placebo three times a day for 16 weeks. If there is no significant outcome obtained between two arms in 16 weeks, placebo will continue until 24 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effects of metformin to prevent frailty in pre-frail non-diabetic elderly. Several outcomes measured in this study are frailty status, quality of life, handgrip strength, gait speed, and serum myostatin levels.

We hypothesize that metformin for 16 weeks could prevent frailty in pre-frail elderly.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-frail elderly;
2. Capable to understand and carry-out the instruction.

Exclusion Criteria:

1. Unwilling to join the study;
2. Diabetes mellitus (oral glucose tolerance test);
3. Abbreviated Mental Test (AMT) score < 8;
4. Geriatric Depression Scale (GDS) score >= 10;
5. Body mass index (BMI) <18,5 Kg/m2;
6. Malnutrition (according to Mini Nutritional Assessment/MNA);
7. Liver cirrhosis, severe liver dysfunction, or serum ALT levels >3 times upper normal limit;
8. Acute illness during inclusion period, eg. pneumonia, pain due to acute arthritis (visual analog scale >6/10), stroke attack, crisis hypertension;
9. Severe cardiac dysfunction: acute decompensated heart failure and/or chronic heart failure functional class III or IV (New York Heart Association classification);
10. Severe pulmonary dysfunction: acute exacerbation of chronic obstructive lung disease stage III or IV (GOLD classification), and/or PaO2 levels < 60 mmHg;
11. Allergy to metformin.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in frailty status at 16 weeks | Baseline and at 16 weeks
  Measurement: Frailty Index 40 items

SECONDARY OUTCOMES:
Change from baseline in health-related quality of life (HrQoL) at 16 weeks | Baseline and at 16 weeks
  Measurement: EQ-5D (with permission)
Change from baseline in handgrip strength at 16 weeks | Baseline and at 16 weeks
  Measurement: handgrip dynamometer (Jamar Hydraulic Hand Dynamometer Model J00105)
Change from baseline in gait speed at 16 weeks | Baseline and at 16 weeks
  Measurement: 15-feet walking test
Change from baseline in serum myostatin levels at 16 weeks | Baseline and at 16 weeks
  Measurement: ELISA test

CONTACTS AND LOCATIONS:
Overall Officials: Purwita Laksmi, MD,SpPD-KGer, Principal Investigator — Division of Geriatrics, Department of Internal Medicine, Universitas Indonesia-Cipto Mangunkusumo General Hospital, Jakarta
Locations (1):
- Cipto Mangunkusumo General Hospital, Central Jakarta, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Sumantri S, Setiati S, Purnamasari D, Dewiasty E. Relationship between metformin and frailty syndrome in elderly people with type 2 diabetes. Acta Med Indones. 2014 Jul;46(3):183-8. PMID 25348180
- [Background] Wang CP, Lorenzo C, Espinoza SE. Frailty Attenuates the Impact of Metformin on Reducing Mortality in Older Adults with Type 2 Diabetes. J Endocrinol Diabetes Obes. 2014;2(2):1031. PMID 25506599